CLINICAL TRIAL: NCT04467177
Title: Efficacy of Oral Glucose in Pain Alleviation Among Healthy Term Neonates Undergoing Circumcision
Brief Title: Analgesic Effect of Oral Glucose in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Amal Naous, Pediatrician, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 18122019
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose group (Experimental): Neonates will receive 30% oral glucose
  Interventions: Other: 30% glucose
- Placebo group (Placebo Comparator): Neonates will receive sterile water
  Interventions: Other: Placebo

INTERVENTIONS:
Other: 30% glucose — Male neonates will receive 2 ml of 30% glucose two minutes prior to circumcision
  Arms: Glucose group
Other: Placebo — Male neonates will receive 2 ml of sterile water two minutes prior to circumcision
  Arms: Placebo group

SUMMARY:
Background: Male circumcision is one of the oldest and most common operations performed all over the world. It can be performed at different ages, using different surgical techniques, for different religious, cultural and medical reasons. It was thought that the newborn baby does not experience pain because of incompletely developed nervous system. However, it has been shown that neurological system known to be associated with pain transmission and modulation, is intact and functional.

OBJECTIVE: Our objective is to determine if a 30% glucose solution would reduce pain after circumcision compared with normal saline.

STUDY DESIGN: This is a randomized placebo-controlled double-blinded clinical trial.

POPULATION: We will include full term neonates, who will be recruited from the inpatient nursery at Makassed General Hospital over a 1-year period.

OUTCOME MEASURE: The primary outcome is to assess efficacy of 30% glucose on pain measured using the Neonatal Infant Pain Score.

Secondary outcome is to assess effect of 30% glucose oh physiologic parameters

ELIGIBILITY:
Inclusion Criteria:

* Estimated gestational age: 37 weeks-42 weeks
* Birth weight: 2500 grams-4000 grams
* Apgar scores a minimum of 7 at 1 and 5 minutes respectively
* Heart rate between 100 and 160 per minutes
* Blood O2 saturation of at least 95%
* No recognized congenital abnormalities

Exclusion Criteria:

* They were transferred to the neonatal intensive care unit (NICU)
* They required respiratory support

Ages: 1 Day to 28 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pain score | Pain will be assessed 1 minute before the procedure and during the procedure
  Pain response will be assessed utilizing the Neonatal Infant Pain Scale. The total pain score ranges from 0 to 10. Scores less than or equal to 3 indicate no pain while scores greater than 3 indicate pain.

SECONDARY OUTCOMES:
Heart rate | 2 minutes before the procedure, during the procedure and one minute after the procedure
  Heart rate (beats per minute) will be recorded
Respiratory rate | 2 minutes before the procedure, during the procedure and one minute after the procedure
  Respiratory rate (breaths per minute) will be recorded
Oxygen saturation | 2 minutes before the procedure, during the procedure and one minute after the procedure
  Oxygen saturation (in percent) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amal Naous, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon